CLINICAL TRIAL: NCT01744938
Title: Preoperative Biliary Drainage for the Lower Malignant Obstructive Jaundice: A Phase III, Randomized, Controlled, Single Center Study.
Brief Title: Preoperative Biliary Drainage for the Lower Malignant Obstructive Jaundice
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIH-STQ-201205001
Record Dates: First submitted 2012-12-05; First posted 2012-12-07 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2012-05

CONDITIONS: Postoperative Complications
Keywords: Postoperative Complications,; mortality,; length of Stay,; economics
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- early surgery (No Intervention): only receiving pancreaticoduodenectomy without preoperative biliary drainage
- preoperative biliary drainage (Experimental): percutaneous preoperative biliary drainage before pancreaticoduodenectomy guided by CT scan
  Interventions: Procedure: preoperative biliary drainage

INTERVENTIONS:
Procedure: preoperative biliary drainage — percutaneous preoperative biliary drainage guided by CT
  Arms: preoperative biliary drainage

SUMMARY:
Patients with the lower malignant obstructive jaundice planned to do the pancreaticoduodenectomy, receiving preoperative biliary drainage or early surgery (without preoperative biliary drainage), both groups has the similar surgical morbidity, no statistics significance.

DETAILED DESCRIPTION:
Patients with the lower malignant obstructive jaundice divided into two groups:early surgery, preoperative biliary drainage + surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the lower malignant obstructive jaundice
* Total bilirubin: 150-350 umol/L

Exclusion Criteria:

* age less than 18
* emergency operation
* biliary tract stent placed
* past history of operation on pancreas
* intraoperative unresectable tumor with pancreaticoduodenectomy
* unresectable tumor or potential resectable tumor with pancreaticoduodenectomy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2012-09; Primary Completion 2016-11 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
the difference in postoperative morbidity | 12 weeks postoperation
  the difference in postoperative morbidity between two groups (preoperative biliary drainage or early surgery (without preoperative biliary drainage))

CONTACTS AND LOCATIONS:
Overall Officials: Song Tian qiang, doctor, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital

REFERENCES:
- [Background] Mumtaz K, Hamid S, Jafri W. Endoscopic retrograde cholangiopancreaticography with or without stenting in patients with pancreaticobiliary malignancy, prior to surgery. Cochrane Database Syst Rev. 2007 Jul 18;2007(3):CD006001. doi: 10.1002/14651858.CD006001.pub2. PMID 17636818
- [Result] van der Gaag NA, Rauws EA, van Eijck CH, Bruno MJ, van der Harst E, Kubben FJ, Gerritsen JJ, Greve JW, Gerhards MF, de Hingh IH, Klinkenbijl JH, Nio CY, de Castro SM, Busch OR, van Gulik TM, Bossuyt PM, Gouma DJ. Preoperative biliary drainage for cancer of the head of the pancreas. N Engl J Med. 2010 Jan 14;362(2):129-37. doi: 10.1056/NEJMoa0903230. PMID 20071702
- [Result] Sewnath ME, Karsten TM, Prins MH, Rauws EJ, Obertop H, Gouma DJ. A meta-analysis on the efficacy of preoperative biliary drainage for tumors causing obstructive jaundice. Ann Surg. 2002 Jul;236(1):17-27. doi: 10.1097/00000658-200207000-00005. PMID 12131081
- [Result] Saleh MM, Norregaard P, Jorgensen HL, Andersen PK, Matzen P. Preoperative endoscopic stent placement before pancreaticoduodenectomy: a meta-analysis of the effect on morbidity and mortality. Gastrointest Endosc. 2002 Oct;56(4):529-34. doi: 10.1067/mge.2002.128161. PMID 12297769
- [Result] Wang Q, Gurusamy KS, Lin H, Xie X, Wang C. Preoperative biliary drainage for obstructive jaundice. Cochrane Database Syst Rev. 2008 Jul 16;(3):CD005444. doi: 10.1002/14651858.CD005444.pub2. PMID 18677779
- [Result] van der Gaag NA, de Castro SM, Rauws EA, Bruno MJ, van Eijck CH, Kuipers EJ, Gerritsen JJ, Rutten JP, Greve JW, Hesselink EJ, Klinkenbijl JH, Rinkes IH, Boerma D, Bonsing BA, van Laarhoven CJ, Kubben FJ, van der Harst E, Sosef MN, Bosscha K, de Hingh IH, Th de Wit L, van Delden OM, Busch OR, van Gulik TM, Bossuyt PM, Gouma DJ. Preoperative biliary drainage for periampullary tumors causing obstructive jaundice; DRainage vs. (direct) OPeration (DROP-trial). BMC Surg. 2007 Mar 12;7:3. doi: 10.1186/1471-2482-7-3. PMID 17352805
- [Result] Tomazic A, Pleskovic A. Surgical outcome after pancreatoduodenectomy: effect of preoperative biliary drainage. Hepatogastroenterology. 2006 Nov-Dec;53(72):944-6. PMID 17153458
- [Result] Pisters PW, Hudec WA, Hess KR, Lee JE, Vauthey JN, Lahoti S, Raijman I, Evans DB. Effect of preoperative biliary decompression on pancreaticoduodenectomy-associated morbidity in 300 consecutive patients. Ann Surg. 2001 Jul;234(1):47-55. doi: 10.1097/00000658-200107000-00008. PMID 11420482
- [Result] van der Gaag NA, Kloek JJ, de Castro SM, Busch OR, van Gulik TM, Gouma DJ. Preoperative biliary drainage in patients with obstructive jaundice: history and current status. J Gastrointest Surg. 2009 Apr;13(4):814-20. doi: 10.1007/s11605-008-0618-4. Epub 2008 Aug 23. PMID 18726134
- [Result] Garcea G, Chee W, Ong SL, Maddern GJ. Preoperative biliary drainage for distal obstruction: the case against revisited. Pancreas. 2010 Mar;39(2):119-26. doi: 10.1097/MPA.0b013e3181bd65de. PMID 19940799
- See also: Tianjin Medical University Cancer Institute and Hospital — http://www.tjmuch.com/